CLINICAL TRIAL: NCT06992609
Title: A Phase IIIb Study of Durvalumab as Consolidation Treatment for Patients Diagnosed With Limited Stage Small Cell Lung Cancer Who Have Not Progressed Following Definitive Concurrent or Sequential Platinum-based Chemoradiation Therapy in Spain (ALBORAN).
Brief Title: Durvalumab After Chemoradiotherapy in Limited Stage Small Cell Lung Cancer.
Acronym: ALBORAN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D419QL00009; 2025-521340-37-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2025-05-12; First posted 2025-05-28 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab (Experimental): Durvalumab after completion of CRT
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — Durvalumab (IV) every 4 weeks until a maximum of 24 months.
  Other Names: Consolidation treatment

SUMMARY:
Lung cancer is a highly prevalent disease worldwide in women and men. In 2022, lung cancer stood as the most frequently diagnosed cancer with approximately 2.48 million new cases on a global scale, followed by cancers of the female breast (11.6%), colorectum (9.6%), prostate (7.3%), and stomach (4.9%).

Lung cancer is the leading cause of cancer death worldwide according to data provided by the International Agency for Research on Cancer. In 2022 they estimated a 1.8 million deaths across the world. Specifically in Spain, from 1980 to 2022, lung cancer led to 745,182 deaths.

Histologically, lung cancer (LC) can be classified into two major subtypes: non-small cell lung cancer (NSCLC) and small cell lung cancer (SCLC), accounting for 85% and 15% of LC patients, respectively. Smoking is the major risk factor for SCLC.

There are two stages of SCLC: limited-stage SCLC (LS-SCLC) and extensive-stage SCLC (ES-SCLC). Limited-stage (LS) means that the cancer is located on the ipsilateral hemithorax that can be encompassed within a radiation port while extensive-stage (ES) means that the cancer has spread widely throughout the lungs, to non-regional lymph nodes or to other organs. At present, LS is identified in ~30% of patients, and ES is identified in ~70% of patients with SCLC.

With a 5-year survival rate of less than 7%, SCLC is still one of the most lethal malignancies and it is also characterized by early metastatic spread. Reflecting this high metastatic capacity, two thirds of patients already have tumor cell dissemination outside the chest at the time of initial diagnosis (ES-SCLC). Therefore, the number of patients with LS-SCLC who can benefit from multimodality therapy with potentially curative intent is limited. SCLC is a highly aggressive form of LC that typically recurs and progresses rapidly despite initial response to chemotherapy and radiotherapy in patients with LS-SCLC.

The etoposide/platinum (EP) combination was the standard of care (SoC) for patients with ES-SCLC until 2019, when the addition of immunotherapy to EP chemotherapy was shown to improve survival, with up to 17% of patients remaining alive at 3 years. On the other hand, the SoC for patients with LS-SCLC is concurrent platinum-based chemoradiotherapy (cCRT) ± prophylactic cranial irradiation (PCI) that remained unchanged for decades. Several studies have shown that concurrent chemoradiotherapy (cCRT) is more effective than sequential CRT (sCRT) in LS-SCLC. Nonetheless, subject to the lymph node regions involvement and treatment-related toxicities, some patients do not undergo concurrent CRT and instead receive sequential CRT. In a non-interventional, retrospective cohort study of limited-stage SCLC patients conducted in France, Italy and the UK, sequential chemoradiotherapy accounts for 37.6% of all treatment patterns while concurrent chemoradiotherapy accounts for 35.1% of the whole therapies used as first line.

ADRIATIC (NCT03703297) is a phase 3, randomized, double-blind, placebo-controlled, multicenter, global study evaluating durvalumab ± tremelimumab as consolidation therapy for patients with LS-SCLC who have not progressed after cCRT. Positive high-level results of the ADRIATIC clinical trial showed durvalumab demonstrated a statistically significant and clinically meaningful improvement in the dual primary endpoints of overall survival (OS) and progression-free survival (PFS) in patients with LS-SCLC who had not progressed following cCRT compared to placebo. Durvalumab was well tolerated, and AEs were consistent with the known safety profile. These data support the consolidation of durvalumab as a new SoC for patients with LS-SCLC who have not progressed after cCRT.

There is limited information on the effectiveness and safety of durvalumab in a broader patient population with LS-SCLC, including those who received sequential CRT.

Therefore, there remains an unmet need for additional data to help support and inform the healthcare decisions on the use of durvalumab as consolidation treatment for patients with LS-SCLC in real-world clinical practice. In addition, ADRIATIC study did not allow to include patients with ECOG PS 2 assessed after CRT.

The present phase IIIb study will assess the safety and effectiveness of durvalumab in real world like LS-SCLC population. Furthermore, this trial will focus on patient characteristics, treatment exposure, administration, quality of life (QoL), effectiveness and safety providing insights into durvalumab use.

DETAILED DESCRIPTION:
Lung cancer is a highly prevalent disease worldwide in women and men. In 2022, lung cancer stood as the most frequently diagnosed cancer with approximately 2.48 million new cases on a global scale, followed by cancers of the female breast (11.6%), colorectum (9.6%), prostate (7.3%), and stomach (4.9%).

Lung cancer is the leading cause of cancer death worldwide according to data provided by the International Agency for Research on Cancer. In 2022 they estimated a 1.8 million deaths across the world. Specifically in Spain, from 1980 to 2022, lung cancer led to 745,182 deaths.

Histologically, lung cancer (LC) can be classified into two major subtypes: non-small cell lung cancer and small cell lung cancer (SCLC), accounting for 85% and 15% of LC patients, respectively. Smoking is the major risk factor for SCLC.

Small cell lung cancer (SCLC) represents approximately 14% of all newly diagnosed lung cancers. SCLC is perhaps the most aggressive form of the disease, distinguishable from non-small-cell lung cancer (NSCLC) by its rapid doubling time, high growth fraction, and early dissemination. It is strongly associated with tobacco smoking and is also associated with an extremely high mutation rate. Moreover, inactivation of TP53 and RB1 occurs frequently, and in a recent study in which sequencing of SCLC tumors was carried out, recurrent mutations were identified in the CREBBP, EP300, and MLL genes that encode histone modifiers. Furthermore, mutations in PTEN, SLIT2, and EPHA7 (as well as focal amplifications of the FGFR1 tyrosine kinase gene) were also observed.

A 2-stage system dividing patients into limited and extensive disease was developed in 1973 by the United States (US) Veteran´s Administration Lung Cancer Study Group. Limited stage was defined as tumor tissue that could be encompassed in a single radiation port, and extensive-stage (ES) disease was defined as any tumor that extended beyond the boundaries of a single radiation port. At present, limited stage is identified in ~30% of patients, and ES is identified in ~70% of patients.

The SoC treatment for LS-SCLC is thoracic radiotherapy (once daily with a total dose of 60 to 66 Gy or twice daily with a total dose of 45 Gy) combined with 4 cycles of either cisplatin or carboplatin and etoposide chemotherapy. In addition, data suggest that prophylactic cranial irradiation (PCI; for patients that respond to initial therapy) may increase the OS and PFS in LS-SCLC patients. Response rates for concurrent CRT in LS-SCLC are approximately 90%, but the majority of patients eventually progress, with median PFS of 10 to 15 months and median OS of 15 to 30 months. Therefore, there is still a significant unmet medical need for additional treatment options for this patient population to improve PFS and OS.

Currently, the 5-year survival rate is approximately 20%-25% for LS-SCLC and barely 1%-2% for ES-SCLC, making SCLC one of the deadliest cancers.

SCLC may be particularly susceptible to immune checkpoint inhibitor therapy given the high mutational burden of this disease. Several recent studies analysing data from different tumor types have demonstrated a correlation between mutational burden and response to checkpoint inhibitors targeting both PD-1 and CTLA-4.

ADRIATIC (NCT03703297) is a phase 3, randomized, double-blind, placebo-controlled, multicenter, global study evaluating durvalumab ± tremelimumab as consolidation therapy for patients with LS-SCLC who have not progressed after cCRT. Positive high-level results of the ADRIATIC clinical trial showed durvalumab demonstrated a statistically significant and clinically meaningful improvement in the dual primary endpoints of overall survival (OS) and progression-free survival (PFS) in patients with LS-SCLC who had not progressed following cCRT compared to placebo. Durvalumab was well tolerated, and AEs were consistent with the known safety profile. These data support the consolidation of durvalumab as a new SoC for patients with LS-SCLC who have not progressed after cCRT.

There is limited information on the effectiveness and safety of durvalumab in a broader patient population with LS-SCLC, including those who received sequential CRT.

The present phase IIIb study will assess the safety and effectiveness of durvalumab in real world LS-SCLC population. Furthermore, the study will focus on patient characteristics, treatment exposure, administration and quality of life (QoL), among others, providing insights into durvalumab use.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients aged ≥18 years at the time of signing the Informed Consent Form (ICF).
* Written informed consent obtained from the patient/legal representative prior to performing any protocol-related procedures. Additionally, signed and dated written genetic and/or biomarker informed consents, respectively, to collect baseline tissue and blood samples for future translational biomarker assessment at baseline, at the initiation of durvalumab maintenance treatment (cycles 1, 2, 3, 4, 7, 10, 13, 19, 26), and at end of treatment/progression.
* Patients must have histologically or cytologically documented limited stage SCLC (stage I-III SCLC [T any, N any, M0] according to the AJCC Cancer Staging Manual, [8th Edition] or the IASLC Staging Manual in Thoracic Oncology [2016]), i.e., patients whose disease can be encompassed within a radical radiation portal. Patients who are stage I or II must be medically inoperable as determined by investigator.
* WHO/ECOG PS of 0, 1 or 2 at enrolment, after CRT. A maximum of 20% of patients with ECOG 2 is allowed.
* Received an appropriate first-line concurrent or sequential chemoradiotherapy regimen as defined below, unless after consultation with the study medical team an alternative is acceptable:

  * Received 3-4 cycles of platinum-based chemotherapy concurrent or sequential with radiotherapy, which must be completed within 1 to 90 days prior to the first dose of durvalumab.
  * The chemotherapy regimen must contain platinum and IV etoposide, administered as per local SoC regimens.
* Received a total dose of radiation of 60 to 66 Gy (±10%) over approximately 6 weeks for standard QD radiation schedules or 45 Gy (±10%) over approximately 3 weeks for hyperfractionated BID radiation schedules.
* Patients must have achieved CR, PR, or SD and not have progressed following definitive, platinum-based chemoradiotherapy. NOTE: PCI may be delivered at the discretion of investigator and local standard of care and must be conducted after the end of CRT and completed between 1 to 90 days to first dose of IP.
* Adequate organ and marrow function (independent of transfusion, infusion, or growth factor support for at least 14 days prior to obtaining screening labs), defined as below:

  * Haemoglobin ≥9.0 g/dL
  * Absolute neutrophil count ≥1.5 x 109/L
  * Platelet count ≥100 x 109/L
  * Serum bilirubin ≤1.5 x the ULN. This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia [predominantly unconjugated bilirubin] in the absence of evidence of hemolysis or hepatic pathology), who will be allowed in consultation with their physician.
  * ALT and AST ≤2.5 x ULN
  * Measured creatinine clearance (CL) >40 mL/min or calculated CL >40 mL/min as determined by Cockcroft-Gault (using actual body weight) Males Creatinine CL (mL/min) = (Weight (kg)×(140-Age))/(72×serum creatinine (mg/dL)) Females Creatinine CL (mL/min) = (Weight (kg)×(140-Age))/(72×serum creatinine (mg/dL) )× 0.85
* Must have a life expectancy of at least 12 weeks.
* Body weight >30 kg.

Exclusion Criteria:

* Mixed SCLC and NSCLC histology.
* Extensive-stage SCLC.
* Any history of grade ≥2 pneumonitis.
* History of allogeneic organ transplantation.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [except for diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis], Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc. The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia.
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement.
  * Any chronic skin condition that does not require systemic therapy.
  * Patients without active disease in the last 5 years may be included but only after consultation with the study physician.
  * Patients with celiac disease controlled by diet alone.
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, active ILD, serious chronic GI conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirements, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of durvalumab and of low potential risk for recurrence.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated carcinoma in situ without evidence of disease.
* History of leptomeningeal carcinomatosis.
* History of active primary immunodeficiency.
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice), hepatitis B (known positive HBsAg result), hepatitis C (HCV), or human immunodeficiency virus (positive HIV 1/2 antibodies).

  * NOTE: Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody and absence of HBsAg) are eligible. Patients positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Any unresolved toxicity NCI Common Terminology Criteria for Adverse Events (CTCAE) Grade ≥2 from previous CRT except for alopecia, vitiligo, and the laboratory values defined in the inclusion criteria:

  * Patients with grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the study physician.
  * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the study physician.
* Brain metastases or spinal cord compression. All patients will have an MRI (preferred) or CT, preferably with IV contrast of the brain, prior to study entry, after CRT.
* Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart).
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
* Patients whose conditions have progressed while on CRT.
* Major surgical procedure (as defined by the Investigator) within 42 days prior to the first dose of IP.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra articular injection).
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent.
  * Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication).
* Participation in another clinical study with an investigational product administered in the last 4 weeks.
* Concurrent enrolment in another clinical study unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
* Female patients who are pregnant or breastfeeding and male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 3 months after the last dose of durvalumab.
* Judgment by the investigator that the patient should not participate in the study because the patient is unlikely to comply with study procedures, restrictions, and requirements.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
To describe the safety profile of durvalumab for patients with LS-SCLC who have not progressed following CRT. | 90 days after last dose of durvalumab of the last patient.
  * Incidence of grade ≥ 3 AEs
  * Incidence of imAE, defined as an AE that is associated with drug exposure and is consistent with an immune-mediated mechanism of action and there is no clear alternate etiology.
  * Incidence of AEs that lead to treatment delays/interruptions or permanent discontinuation.

SECONDARY OUTCOMES:
To describe effectiveness of durvalumab for patients with LS-SCLC who have not progressed following CRT. | From the date of first dose of durvalumab until the date of disease progression, death, withdrawn from study, or end of study (approximately 56 months)
  • Progression-Free Survival (PFS). Progression-Free Survival defined as the time from the date of first dose of durvalumab until the date of objective disease progression according RECIST 1.1 criteria assessed by investigator, or death (by any cause in the absence of progression). The measure of interest is the median PFS.
To describe effectiveness of durvalumab for patients with LS-SCLC who have not progressed following CRT. | Up to 36 months
  • Overall Survival (OS) rate at 36 months, defined as the percentage of patients that are still alive at 36 months.
To further describe safety profile of durvalumab for patients with LS-SCLC who have not progressed following CRT. | 90 days after last dose of durvalumab of the last patient.
  * All AEs.
  * Serious AEs.

CONTACTS AND LOCATIONS:
Locations (12):
- Spain (12):
  - Research Site, A Coruña
  - Research Site, Badajoz
  - Research Site, Barakaldo
  - Research Site, Barcelona
  - Research Site, Jerez de la Frontera
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Oviedo
  - Research Site, Santander
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/